CLINICAL TRIAL: NCT00654303
Title: ZD4522 Long Term Extension Trial
Brief Title: OLE Study to Evaluate Safety / Efficacy of ZD4522
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Elisabeth Björk, AstraZeneca
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4522IL/0034; D3560C00034
Record Dates: First submitted 2008-04-02; First posted 2008-04-07 (Estimated); Last update posted 2009-03-16 (Estimated); Status verified 2009-03

CONDITIONS: Hypercholesterolaemia
Keywords: Cholesterol; Hypercholesterolaemia; Statins
MeSH Terms: conditions — Hypercholesterolemia | interventions — Rosuvastatin Calcium

ARMS (1):
- 1 (Experimental): Rosuvastatin
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin
  Other Names: Crestor

SUMMARY:
The purpose of this study is to assess the long term safety of Crestor.

ELIGIBILITY:
Inclusion Criteria:

* Completion of previous Crestor study as listed in the protocol.

Exclusion Criteria:

* Pregnant or breast feeding women, or not using appropriate contraception.
* Abnormal lab values as listed in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3500 (Estimated)
Dates: Start 1999-08; Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Safety, as determined by adverse events, laboratory data, physical examination and ECG. | 12 weekly

SECONDARY OUTCOMES:
Success in achieving goals for Cholesterol levels | 12 weekly

CONTACTS AND LOCATIONS:
Overall Officials: Elinor Miller, MD, Study Director — AstraZeneca